CLINICAL TRIAL: NCT05312983
Title: Development of a Battery of Audiological Tests for the Precision Diagnosis of Age-related Hearing Loss
Acronym: AUDIOGENAGE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Pasteur (Industry)
Collaborators: CEntre de Recherche et d'Innovation en Audiologie Humaine (Unknown); Laboratoire de correction auditive (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2021-062; 2021-A02543-38 (Other: ID-RCB)
Record Dates: First submitted 2022-02-25; First posted 2022-04-06 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Presbyacusis
Keywords: presbyacusis; aging; audiology; genetic
MeSH Terms: conditions — Presbycusis | interventions — Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: 2 groups :
  * 500 participants with early onset presbycusis
  * 200 participants with normal hearing for their age
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- people over the age of 18 who agree to participate in the research. (Experimental): They are either people who have a hearing loss about 20 years older than their age and wear a hearing aid (or come in for a hearing aid), or people over the age of 40 with normal hearing for their age.
  Interventions: Other: Audiological and vestibular tests; Other: Blood sampling; Other: neurocognitive self-questionnaire

INTERVENTIONS:
Other: Audiological and vestibular tests — 6h of audiological and vestibular tests divide in 3 sessions :
  * Session A : objective audiological tests
  * Session B ; subjective audiological tests
  * Session C : balance tests.
Other: Blood sampling — A 10 mL blood sample will be collected during the study.
Other: neurocognitive self-questionnaire — Four self-questionnaires to fill out to measure sleep quality, memory and emotional state

SUMMARY:
Age-related hearing loss, or presbycusis, is caused by many genetic and environmental factors. Its prevalence poses a public health challenge of early identification and effective hearing aid treatment. However, the lack of screening and of a validated audiological test battery to diagnose an individual's needs and to guide hearing aid adjustments is a major obstacle.

Furthermore, monogenic forms of hearing loss affect only one functional module of hearing. The audiological test(s) dependent on the function of this module are affected, in a progressive manner, but not the others. A previous study showed that in early onset presbycusis patients, a quarter of the subjects tested were affected by monogenic presbycusis.

The collection of audiological and vestibular tests, carried out on proven monogenic presbycusis patients and compared to that of normal hearing patients, would constitute a battery of tests allowing a precision diagnosis, then developed to all forms of presbycusis in order to study if the identification of abnormal functional modules can usefully guide the diagnosis and the early fitting.

DETAILED DESCRIPTION:
The AUDIOGENAGE project is a multi-center, non-invasive case-control study conducted by CERIAH (CEntre de Recherche et d'Innovation en Human Audiology) and LCA (Laboratory de correction auditive) in 700 volunteer participants identified in two groups:

* 500 Patients with age-related hearing loss of anticipated onset,
* 200 Control subjects, considered as normal hearing for their age at inclusion.

All participants will undergo 6h audiological and vestibular tests, and also neurocognitive test (self-questionnaire). These tests will be conducted over 2 to 4 visits. A 10 mL-blood sample will be collected for a genetic analysis.

ELIGIBILITY:
Inclusion Criteria:

For all participants:

* Be over the age of 18,
* Be affiliated to a social security system,
* Have a good command of the French language (oral and written).

For the group of participants with anticipated presbycusis:

* Over the age of 40, having a hearing aid recipient or coming for a first hearing aid recipient
* Between 18 and 40, having a hearing aid recipient, coming for a first hearing aid recipient or declare a progressive genetic birth defect

For healthy volunteers:

- Have no known hearing loss.

Exclusion Criteria:

* Report having been chronically exposed to loud sounds.
* Have a history of ototoxic substances,
* To have sequelae of ear infections and/or a history of ENT disease that permanently affects hearing or balance,
* Have an ethnic origin for which the Pasteur Institute does not have information on the frequency of variants of the genes studied.
* Have type II diabetes,
* Have a neurological or psychiatric condition that interferes with comprehension or ability to move,
* Be under guardianship,
* Be deprived of liberty by judicial or administrative decision, or be subject to legal protection,
* Not being subject to a social security system,
* Taking narcotic substances, alcohol or medication that diminishes cognitive abilities.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 700 (Estimated)
Dates: Start 2022-07-28 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Measurement of specificity and sensitivity of the audiological test battery in participants with early-onset presbycusis after identification of pathogenic variants by sequencing and division into subgroups. | 2 years
  specifity and sensitivity will be calculated to identify which tests or combinations of audiological and vestibular tests will be the most discriminating in characterizing each functional module of hearing from participants with monogenic forms of presbycusis of anticipated onset, each affecting a determined functional module, in comparison with an age-matched control group.

SECONDARY OUTCOMES:
Normative values for audiological and vestibular tests will be determined | 4 years and 6 months
  Measurement of values by age range for all audiological and vestibular tests from the results of participants in the control group
Whole-exome sequencing of samples from participants with non-monogenic presbycusis | 4 years and 6 months
  Whole-exome sequencing will be performed to establish a list of new candidate genes for predisposition to presbycusis.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Avan, MD, Principal Investigator — CERIAH
Locations (2):
- France (2):
  - Laboratoire de correction auditive, Paris
  - CEntre de Recherche et d'Innovation en Audiologie Humaine, Paris